CLINICAL TRIAL: NCT00985491
Title: A Pilot Trial of the GI EndoBarrier Liner for Short Term Weight Loss in Subjects Who Are Candidates for Bariatric Surgery
Brief Title: Study for Short Term Weight Loss in Candidates for Bariatric Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-1
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device (Experimental): All patients will be implanted with the Endobarrier Liner device.
  Interventions: Device: Endobarrier Liner

INTERVENTIONS:
Device: Endobarrier Liner — Medical device placed endoscopically in the duodenum
  Other Names: GI Sleeve

SUMMARY:
The purpose of this study is to determine whether the GI Endobarrier Liner is safe and effective.

DETAILED DESCRIPTION:
Patients with obesity are at significantly greater risk of developing significant co-morbid complications, and are associated with an increased risk in all-cause mortality. The GI Endobarrier Liner represents a viable alternative to other short-term weight loss methods. It is a minimally invasive endoscopic procedure, which may allow patients to recover faster with less morbidity and mortality. This study is investigating the safety and efficacy of the GI Endobarrier Liner in patients who are candidates for bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 55 years - Male or Female
* BMI > 35 with significant comorbidities (i.e. hypertension, or hyperlipidemia, or diabetes) or > 40 BMI <60 (with or without a co-morbid condition)
* History of failure with nonsurgical weight loss methods
* Candidates for Roux-en-Y gastric bypass
* Willing to comply with trial requirements
* Signed an ICF
* Post-menopausal women with surgical sterilization or following any treatment or family planning and not planning to become pregnant during the course of the investigation

Exclusion Criteria:

* Treatment represents an unreasonable risk to the subject
* Pregnant or have intention of becoming pregnant for the duration of the trial
* Unresolved alcohol or drug addiction
* Receiving weight loss medications (prescription, over-the-counter, or herbal dietary medications)
* Previous gastrointestinal surgery that could affect the ability to place the EndoBarrier Liner or the function of the implant
* Active GERD
* Symptomatic kidney stones prior to implant
* Iron deficiency and/or iron deficiency anemia
* History of Inflammatory bowel disease or condition of the gastrointestinal tract, such as ulcers or Crohn's disease
* Symptomatic gallstones prior to implant
* Symptomatic coronary artery disease or pulmonary dysfunction
* Known infection at the time of implant
* History of congenital or acquired anomalies of the gastrointestinal tract such as atresias or stenoses
* Pancreatitis or other serious organic conditions
* Requiring prescription anticoagulation therapy
* Unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during the implant period
* Having or Family history of a known diagnosis or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
* Participating in another ongoing investigational clinical trial
* Mentally retarded or emotionally unstable, or exhibits psychological characteristics requiring medication that affects appetite (i.e. tricyclic antidepressants and atypical antipsychotic medications) which, in the opinion of the Investigator, makes the subject a poor candidate for device placement or clinical trial
* Active Helicobacter pylori (Note: Subjects may be enrolled if they had a prior history of H. Pylori and were successfully treated)
* Having or a history of coagulopathy, upper gastro-intestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2008-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex P Escalona, MD, Principal Investigator — Pontificia Universidad Catolica de Chile, Santiago, Chile
Locations (1):
- Dr. Nicholas Quezada, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Escalona A, Pimentel F, Sharp A, Becerra P, Slako M, Turiel D, Munoz R, Bambs C, Guzman S, Ibanez L, Gersin K. Weight loss and metabolic improvement in morbidly obese subjects implanted for 1 year with an endoscopic duodenal-jejunal bypass liner. Ann Surg. 2012 Jun;255(6):1080-5. doi: 10.1097/SLA.0b013e31825498c4. PMID 22534421

RESULTS

PARTICIPANT FLOW:
Groups:
- EndoBarrier Liner Device: All patients will be implanted with the Endobarrier Liner device.
  Endobarrier Liner: Medical device placed endoscopically in the duodenum
Period: Overall Study
Arm/Group | EndoBarrier Liner Device
Started | 46 (46 subjects underwent an attempted implantation procedure)
Received Device | 43
Completed | 27 (43 subjects received a device, 27 subjects completed 12 month implant period)
Not Completed | 19
Not completed — Adverse Event | 8
Not completed — device migration | 7
Not completed — Withdrawal by Subject | 1
Not completed — implant failure | 3

BASELINE CHARACTERISTICS:
Groups:
- EndoBarrier Liner Device: 46 subjects were enrolled. 3 subjects were implant failures. 43 Subjects received the device.
  Endobarrier Liner: Medical device placed endoscopically in the duodenum
Arm/Group | EndoBarrier Liner Device
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 10
Region of Enrollment [Number; unit: participants]
  Chile | 43
HbA1c [Mean (Standard Deviation); unit: %] | 7.7 (2.03)
Baseline Weight [Mean (Standard Deviation); unit: kg] | 110.3 (18.52)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of % Excess Weight Loss
Description: Primary efficacy was assessment of the percent excess weight loss (%EWL) at Week 52 or last assessment. Excess weight was determined from ideal body weights based on a body mass index (BMI) of 25 kg/m2. Percent excess weight loss from baseline to 12 months was calculated as [(baseline weight minus the 12-month weight) / (baseline weight minus the ideal body weight)] * 100).
Time Frame: 12 months
Measure: Mean (Standard Error); unit: %EWL
Arm/Group | EndoBarrier Liner Device
Number analyzed (Participants) | 27
%EWL | 45.4 (20.3)

2. Secondary Outcome: Improvement in Type 2 Diabetic Status
Description: Subjects who achieved HbA1c reduction of 0.5%
Time Frame: 12 months
Population: 7 subjects were enrolled that had Type 2 Diabetes; endpoint evaluated subjects who achieved HbA1c reduction of 0.5%
Measure: Number; unit: % of subjects with T2DM
Arm/Group | Device
Number analyzed (Participants) | 7
% of subjects with T2DM | 57.1

ADVERSE EVENTS:
Arm/Group | EndoBarrier Liner Device
Serious Adverse Events (participants affected / at risk) | 21/46
Other Adverse Events (participants affected / at risk) | 39/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier Liner Device (N=46)
Abdominal pain upper (Gastrointestinal disorders) | 19 (19)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 2 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Endoscopy (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Benign ovarian tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier Liner Device (N=46)
Abdominal pain upper (Gastrointestinal disorders) | 36 (78)
Nausea (Gastrointestinal disorders) | 15 (18)
Vomiting (Gastrointestinal disorders) | 15 (21)
Procedural nausea (Gastrointestinal disorders) | 8 (8)
Procedural vomiting (Injury, poisoning and procedural complications) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No